CLINICAL TRIAL: NCT05705115
Title: A Randomized Study to Investigate Central and Cerebral Hemodynamic Effects and Volume Kinetics of Ringer´s Acetate Compared With no Intravenous Fluids, During Experimental Hypovolemia Compared With Euvolemia, in Healthy Human Volunteers
Brief Title: Acetated Ringer´s Solution in Experimental Hypovolemia
Acronym: Volu-Flow
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Lars Øivind Høiseth, M.D., PhD, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Volu-Flow
Record Dates: First submitted 2023-01-21; First posted 2023-01-30 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Hypovolemia; Fluid Loss; Hemodynamic Instability
MeSH Terms: conditions — Hypovolemia | interventions — Lower Body Negative Pressure

STUDY DESIGN:
Intervention Model Description: * Block randomized
  * Placebo controlled
  * Single center
  * Crossover
  * Factorial 2x2
Masking Description: Open-label using blinded randomization. The intervention to be taken by a participant will be assigned using randomization envelopes, opened at visit 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- LBNP 0 + no intravenous fluid (No Intervention)
- LBNP 0 + Ringer's acetate (Experimental)
  Interventions: Drug: Ringer acetate
- LBNP 40 + no intravenous fluid (Active Comparator)
  Interventions: Other: Lower body negative pressure
- LBNP 40 + Ringer's acetate (Experimental)
  Interventions: Drug: Ringer acetate; Other: Lower body negative pressure

INTERVENTIONS:
Drug: Ringer acetate — Ringer acetate 5 ml/kg.
  Arms: LBNP 0 + Ringer's acetate; LBNP 40 + Ringer's acetate
Other: Lower body negative pressure — Lower body negative pressure, 40 mmHg. Experimental hypovolemia.
  Arms: LBNP 40 + Ringer's acetate; LBNP 40 + no intravenous fluid

SUMMARY:
Intravenous fluids are often given to increase stroke volume and thereby improve global oxygen delivery. The effect is however often transient, but the effect of a fluid bolus on stroke volume and other hemodynamic variables over time are poorly described. The volume effect of a fluid bolus (effect on blood volume) can be calculated by measuring Haemoglobin. The purpose of this study is to elucidate the hemodynamic effects of a fluid bolus during normovolemia and hypovolemia in healthy volunteers. Study details include:

• Study Duration: 2 visits of approximately 2 h duration each + follow-up visit. Visits 1 and 2 are at least 2 days apart. Number of Participants: A maximum of 15 participants will be enrolled to study intervention such that 12 evaluable participants complete the study

DETAILED DESCRIPTION:
Administration of intravenous fluids is one of the most commonly performed procedures in anaesthesia, critical care and emergency medicine. Intravenous fluids can be given to achieve specific goals depending on the type of fluid, but often, fluid is given simply to expand the intravascular volume. The volume-expanding effect of intravenous fluids is however time-dependent, and often of limited duration as fluid is distributed out of the intravascular space and eliminated mainly in the kidneys.

The goal of intravascular volume expansion is to improve haemodynamic variables, such as SV, CO and ABP. The reasoning is that volume expansion increases SV mainly mediated by the Frank-Starling mechanism. The degree to which SV increases with volume expansion is termed fluid responsiveness.1 The increase in SV does however in most cases seem to be transient. The reason for the transient nature of the hemodynamic response is not known, but may be related to reduction in intravascular volume expansion as described above or other factors, such as vasodilation.

Calculation of volume expansion:

The volume-expanding effect of intravenous fluids has been studied by measuring concentration of hemoglobin. Under the assumption that hemoglobin is evenly distributed in, and does not leave the intravascular space, intravascular volume can be calculated and kinetic studies of the volume effect (volume kinetics) can be performed.

Hb = intravascular amount of hemoglobin V0 = Intravascular volume at time 0 Vt = Intravascular volume at time t [Hb]0 = Hemoglobin concentration at time 0 [Hb]t = Hemoglobin concentration at time t Eq1: (Hb)o= Hb/Vo. Vo = Hb/(Hb)o Eq 2: (Hb)t= Hb/Vt. Vo = Hb/(Hb)t.

Assuming that the amount of hemoglobin is constant, from Eq 1 ang Eq 2, it follows that:

Eq 3: Vt/V0=(Hb)o/(Hb)t which therefore gives the relative value of intravascular volume at time=t to compared to time=0; Vt_rel.

Kinetic model of outcomes:

Similar to the volume expansion, the relative value of the hemodynamic variables compared to baseline can be calculated, expressed as value at time=t, Vt.

A pharmacokinetic model can then be fitted to the observations. In a two-compartment model, the relative value (e.g. volume) of the observed value at time=t (Vt) can be described as:

Eq 4: V_(t_rel)=D(〖Ae〗^(-αt)+〖Be〗^(-βt))

A one-compartment model can be described as:

Eq 5: V_(t_rel)=D(〖Ae〗^(-αt)) A two-compartment model will typically describe a rapid equilibration with one compartment and a slower elimination. Initially the reduction in Vt is dominated by distribution, and later by the slower elimination. Each of these effects have their own half-lives, given by α and β. For a one-compartment model, the reduction in Vt is best described by a single half-life.

LBNP-model:

LBNP is a model that has been used for several decades. Lower body negative pressure (LBNP) is a model of central hypovolemia where negative pressure is applied to the body from the waist-down. Thereby, blood is displaced from the central compartment of the upper body to the lower extremities and pelvis. The model has been used for more than half a century and is considered useful model for studying hypovolemia in conscious volunteers.

The volume kinetics of intravenous fluids has been shown to be affected by volume status, with a longer lasting volume effect during hypovolaemia.The effects of volume status on the hemodynamic response to intravenous fluids has been less explored.

Aim of the study The aim of the present study is to explore the effects over time of an intravenous fluid bolus. The effects on the volume expanding effects and the hemodynamic effects will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination and focused cardiac ultrasound
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
* Sex and Contraceptive/Barrier Requirements Male participants: Not applicable. Female participants: Use of adequate birth control for women of childbearing potential.
* A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile when sexually active. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
* Inclusion of WOCBP is possible when either:
* Using at least an acceptable effective contraceptive measure (combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner or sexual abstinence). As a minimum contraception should be maintained until treatment discontinuation. or
* Confirmed negative highly sensitive urine or serum pregnancy test at screening. A pregnancy test is performed at any visit before administering IMP if more than 14 days have passed since last pregnancy test. There will be no demand for post-intervention contraception.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

1. Any medical condition limiting physical exertional capacity or requiring regular medication (allergy and contraceptives excepted).
2. Pregnancy.
3. Breastfeeding.
4. History of syncope (syncope of presumed vasovagal nature with known precipitating factor excepted).
5. Any known cardiac arrhythmia. Prior/Concomitant Therapy
6. Any drug (contraceptives excepted) used on a regular basis for a chronic condition (allergy excepted).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-03-02 (Actual); Primary Completion 2024-07-29 (Estimated); Study Completion 2024-07-29 (Estimated)

PRIMARY OUTCOMES:
Cardiac stroke volume | 120 minutes
  Half-life of change in cardiac stroke volume

SECONDARY OUTCOMES:
Intravascular volume | 120 minutes
  Half-life of change in intravascular volume
Middle cerebral artery blood flow velocity | 120 minutes
  Half-life of change in middle cerebral artery blood flow velocity

OTHER OUTCOMES:
Hemodynamic response | 120 minutes
  Half-lives of mean arterial pressure, heart rate and cardiac output

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No